CLINICAL TRIAL: NCT00532038
Title: An Open-Label, Long-Term Safety Study to Evaluate the Safety of ThermoProfen™ for the Treatment of Mild to Moderate Pain Associated With Osteoarthritis of the Knee
Brief Title: A Phase 3 Study to Evaluate the Long-Term Safety of ThermoProfen™ in Patients With Mild to Moderate Pain Associated With Osteoarthritis of the Knee.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Corporate decision
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZMK-304
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Pain
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ThermoProfen™ (Matrix Transdermal Ketoprofen/CHADD™ System) — Patients will apply ThermoProfen daily for approximately 12 hours for up to 12 months for treatment of the pain associated with osteoarthritis of the knee.

SUMMARY:
ThermoProfen is a transdermal ketoprofen patch that is integrated with a long-lasting CHADD (Controlled Heat-Assisted Drug Delivery) unit for the treatment of chronic pain associated with osteoarthritis. This study will evaluate the safety of long-term administration of ThermoProfen™ for the pain associated with osteoarthritis of the knee in adults. The study will be conducted in patients with pain associated with osteoarthritis and who have completed a previous efficacy study of ThermoProfen.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the safety of long-term administration of ThermoProfen for the pain associated with osteoarthritis of the knee in adults.

ELIGIBILITY:
Inclusion Criteria:

* Patient completed a previous efficacy study of ThermoProfen.

Exclusion Criteria:

* Patient has a known allergy to nonsteroidal anti-inflammatory drugs (NSAIDs) (including aspirin).
* Patient has a suspected hypersensitivity, allergy, or other contraindication to any compound present in the study medication or has a known sensitivity to adhesive components similar to those used in ThermoProfen (such as that found in adhesive bandages, e.g. Band-Aid®).
* Patient has asthma that has been induced or made worse by the use of aspirin or any other NSAID.
* Patient has a relevant history of serious gastrointestinal disease.
* Patient has a defect, injury, or dermatologic disease or condition on the skin area where the study patch will be applied that may interfere with tolerability or post-application evaluations.
* Patient has neurological or psychiatric disease sufficient to compromise data collection or integrity.
* Patient is taking warfarin, heparin, or low molecular weight heparin.
* Patient, if female, is pregnant or breastfeeding or is of childbearing potential and not practicing adequate birth control.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of long-term administration of ThermoProfen™ | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — ZARS Pharma
Locations (20):
- United States (20):
  - Anaheim, California
  - San Diego, California
  - Westlake Village, California
  - Clearwater, Florida
  - Pembroke Pines, Florida
  - Springfield, Illinois
  - Evansville, Indiana
  - Overland Park, Kansas
  - Baltimore, Maryland
  - Wheaton, Maryland
  - Kansas City, Missouri
  - Mercerville, New Jersey
  - Raleigh, North Carolina
  - Lake Oswego, Oregon
  - Duncansville, Pennsylvania
  - Erie, Pennsylvania
  - Anderson, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas